CLINICAL TRIAL: NCT04694430
Title: A Integration of Respiratory Medicine and Prevention Multi-center Study to Determine the Prevalence and Influence of Pertussis on Chronic Obstructive Pulmonary Disease Exacerbation in Shenzhen by National Respiratory Diseases Clinical Medicine Research Center
Brief Title: A Multi-center Study to Determine the Prevalence and Influence of Pertussis on COPD Exacerbation in Shenzhen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WLW-COPD-Pertussis
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: COPD Exacerbation; Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Throat swab, Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe exacerbation of COPD: N = 250
  Interventions: Procedure: Blood sample; Other: Data collection; Procedure: Throat swab
- Mild and moderate exacerbations of COPD: N = 250
  Interventions: Procedure: Blood sample; Other: Data collection; Procedure: Throat swab

INTERVENTIONS:
Procedure: Blood sample — 2 ml venous blood was collected and separated into serum.
Other: Data collection — 1. Whether the patient has been vaccinated with DPT vaccine and record the time of vaccination;
  2. Medication situation of patients in the past year, including rescue drugs, antitussive and expectorant drugs, inhaled corticosteroids and antibiotics;
  3. Assess COPD using ABCD assessment tool.
Procedure: Throat swab — Before the collection of oropharyngeal swabs, instruct the patient to wash the mouth or gargle, fix the patient's head, open the mouth and expose the throat. If necessary, use a tongue depressor to gently press the tongue.
  Use the swab to wipe the secretion on both sides of the palatal arch, pharynx and tonsil with a sensitive and gentle action, and quickly withdraw the swab to avoid contacting other parts of the mouth.
  Put the swab in the sterile test tube, plug the opening with cotton ball, and send it for inspection and registration in time.

SUMMARY:
A prospective, multi-center, observational clinical trail. Aim to evaluate the real incidence of chronic obstructive pulmonary disease (COPD) pertussis and the impact of pertussis on COPD exacerbation.

DETAILED DESCRIPTION:
1. Investigate the incidence and epidemiological characteristics of pertussis infection in COPD population.
2. To explore the relationship between pertussis infection and COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of acute COPD

Exclusion Criteria:

- Major diseases except COPD; Significant abnormality in laboratory examination; Clinical diagnosis of lung cancer, bronchiectasis, pneumoconiosis or other simple restrictive ventilation dysfunction; Patients with a history of asthma, allergic rhinitis, or a blood eosinophil count of 2600/mm3 (0.6x10^9/L) within 4 weeks; Currently suffering from active tuberculosis; Patients with life-threatening pulmonary embolism, or al-antitrypsin deficiency, or cystic fibrosis; Patients who have undergone lung resection.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute COPD in Shenzhen
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prevalence of pertussis among COPD | Day 0 of each subject at the time of enrollment.
  According to the positive rate of bordetella pertussis nucleic acid, evaluate the prevalence of pertussis in COPD.
Evaluation of the correlation between pertussis and COPD exacerbation | Day 0 of each subject at the time of enrollment.
  Evaluate the correlation between pertussis infection and COPD exacerbation by pertussis positive rate and exacerbation degree.

SECONDARY OUTCOMES:
Evaluation of the seroprevalence of Bordetella pertussis in COPD | Day 0 of each subject at the time of enrollment.
  According to anti-pertussis (anti-PT) antibody levels, assess the overall seroprevalence of Bordetella pertussis in COPD.
Evaluation of the cut-off value for serological diagnosis of pertussis. | Day 0 of each subject at the time of enrollment.
  By comparing the nucleic acid and antibody levels of Bordetella pertussis to evaluate the antibody cut-off value for serological diagnosis of pertussis.
Evaluation of the subtype of bordetella pertussis. | Day 0 of each subject at the time of enrollment.
  According to the level and pattern of different anti-pertussis antibodies (anti-PT, anti-FHA, anti-PRN, anti-FIM2, anti-FIM3), assess the subtype of Bordetella pertussis.

CONTACTS AND LOCATIONS:
Overall Officials: Lingwei Wang, Study Director — Shenzhen People's Hospital
Locations (27):
- China (27):
  - Fuyong people's Hospital of Baoan District, Shenzhen, Shenzhen
  - General Hospital of Shenzhen University, Shenzhen
  - Longhua Branch of Shenzhen People's Hospital, Shenzhen
  - Nanshan District People's Hospital, Shenzhen
  - Peking university shenzhen hospital, Shenzhen
  - Shenzhen Bao'an District Central Hospital, Shenzhen
  - Shenzhen Bao'an District People's Hospital, Shenzhen
  - Shenzhen Hospital of Beijing University of traditional Chinese Medicine, Shenzhen
  - Shenzhen Hospital of Guangzhou University of traditional Chinese Medicine, Shenzhen
  - Shenzhen Hospital of Southern Medical University, Shenzhen
  - Shenzhen Hospital of the University of Hong Kong, Shenzhen
  - Shenzhen Longgang District Central Hospital, Shenzhen
  - Shenzhen Longgang District People's Hospital, Shenzhen
  - Shenzhen Longgang District Second People's Hospital, Shenzhen
  - Shenzhen Longgang District Third People's Hospital, Shenzhen
  - Shenzhen Longhua District Central Hospital, Shenzhen
  - Shenzhen Longhua District People's Hospital, Shenzhen
  - Shenzhen Luohu District People's Hospital, Shenzhen
  - Shenzhen People's Hospital, Shenzhen
  - Shenzhen Pingshan District Hospital of traditional Chinese Medicine, Shenzhen
  - Shenzhen Pingshan District People's Hospital, Shenzhen
  - Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen
  - Shenzhen Second People's Hospital, Shenzhen
  - Shenzhen TCM Hospital, Shenzhen
  - Shenzhen Yantian District People's Hospital, Shenzhen
  - South University of science and Technology Hospital, Shenzhen
  - The eighth Affiliated Hospital of Sun Yat sen University, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manian P. Chronic obstructive pulmonary disease classification, phenotypes and risk assessment. J Thorac Dis. 2019 Sep;11(Suppl 14):S1761-S1766. doi: 10.21037/jtd.2019.05.10. PMID 31632753
- [Background] Santus P, Pecchiari M, Tursi F, Valenti V, Saad M, Radovanovic D. The Airways' Mechanical Stress in Lung Disease: Implications for COPD Pathophysiology and Treatment Evaluation. Can Respir J. 2019 Sep 5;2019:3546056. doi: 10.1155/2019/3546056. eCollection 2019. PMID 31583033
- [Background] Canepa M, Franssen FME, Olschewski H, Lainscak M, Bohm M, Tavazzi L, Rosenkranz S. Diagnostic and Therapeutic Gaps in Patients With Heart Failure and Chronic Obstructive Pulmonary Disease. JACC Heart Fail. 2019 Oct;7(10):823-833. doi: 10.1016/j.jchf.2019.05.009. Epub 2019 Sep 11. PMID 31521680
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Wang M, Luo X, Xu S, Liu W, Ding F, Zhang X, Wang L, Liu J, Hu J, Wang W. Trends in smoking prevalence and implication for chronic diseases in China: serial national cross-sectional surveys from 2003 to 2013. Lancet Respir Med. 2019 Jan;7(1):35-45. doi: 10.1016/S2213-2600(18)30432-6. Epub 2018 Oct 25. PMID 30482646
- [Background] Jia JH, Guo Q, Wan CM. [Resurgence and vaccine strategies of pertussis]. Zhonghua Er Ke Za Zhi. 2020 Aug 2;58(8):686-689. doi: 10.3760/cma.j.cn112140-20200116-00036. Chinese. PMID 32842393
- [Background] Huang H, Zhu T, Gao C, Gao Z, Liu Y, Ding Y, Sun J, Guo L, Liu P, Chen D, Wang L, Wu S, Zhang Y. Epidemiological features of pertussis resurgence based on community populations with high vaccination coverage in China. Epidemiol Infect. 2015 Jul;143(9):1950-6. doi: 10.1017/S095026881400260X. Epub 2014 Oct 7. PMID 25286969
- [Background] Huang HT, Gao ZG, Liu Y, Sun J, Liu P, Wang LJ, Li Y, Zhang J, Zhang Y. [Epidemiology of pertussis in adults and related factors in Tianjin, 2005-2014]. Zhonghua Liu Xing Bing Xue Za Zhi. 2016 May;37(5):678-81. doi: 10.3760/cma.j.issn.0254-6450.2016.05.018. Chinese. PMID 27188361
- [Background] Wang Y, Xu C, Ren J, Zhao Y, Li Y, Wang L, Yao S. The long-term effects of meteorological parameters on pertussis infections in Chongqing, China, 2004-2018. Sci Rep. 2020 Oct 14;10(1):17235. doi: 10.1038/s41598-020-74363-8. PMID 33057239
- [Background] Wang H, Zheng Y, de Groot R, Yang Y, Diavatopoulos DA, Chen Y, de Jonge MI, Deng J. High prevalence of Bordetella pertussis in young hospitalized infants with acute respiratory infection in the south of China: age- and season-dependent effects. J Infect. 2020 May;80(5):578-606. doi: 10.1016/j.jinf.2020.01.009. Epub 2020 Jan 23. No abstract available. PMID 31981637